CLINICAL TRIAL: NCT06835465
Title: A Phase 1, Open-Label, Single-Dose, Two-Period, Fixed Sequence, Crossover Study to Determine the Effect of Rifampin on the Pharmacokinetics of Divarasib in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Rifampin on the Pharmacokinetics of Divarasib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GP45718
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive a single oral dose of Divarasib on Day 1.
  Interventions: Drug: Divarasib
- Treatment B (Experimental): Participants will receive Rifampin once daily (QD) on Days 1 to 7 and Days 9 to 13. Participants will receive Divarasib followed by Rifampin on Day 8.
  Interventions: Drug: Divarasib; Drug: Rifampin

INTERVENTIONS:
Drug: Divarasib — Divarasib will be administered as a single oral dose as specified for the respective period.
Drug: Rifampin — Rifampin will be administered QD on Days 1 to 7 and Days 9 to 13 and as a single oral dose on Day 8 as specified for the respective period.
  Arms: Treatment B

SUMMARY:
This is a phase 1, open-label, two-period, fixed sequence drug-drug interaction study to evaluate the impact of multiple doses of rifampin on the pharmacokinetics (PK) and safety of divarasib in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential
* Within body mass index (BMI) range of 18.0 to 32.0 kg/m2, inclusive

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* Poor peripheral venous access

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Divarasib | Day 1 of Period 1 and Day 8 of Period 2
Area Under the Concentration-time Curve Extrapolated to Infinity (AUC0-inf) of Divarasib | Day 1 of Period 1 and Day 8 of Period 2
Area Under the Concentration-time Curve from Hour 0 to the Last Measurable Concentration (AUC0-t) of Divarasib | Day 1 of Period 1 and Day 8 of Period 2

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Fortrea Dallas CRU, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No